CLINICAL TRIAL: NCT00750724
Title: Phase 3 Study GoON and MRI Improvement in OA Knee
Brief Title: Efficacy Study of "Go On" in Magnetic Resonance Imaging (MRI) Improvement in Osteoarthritis (OA) Knee
Acronym: GoOn MRI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Faculty of Medicine, Department of Orthopedics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Faculty of Medicine, Khon Kaen
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2009-07

CONDITIONS: Osteoarthritis
Keywords: Hyaluronic acid,; OA knee,; MRI
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Placebo Comparator): 2 ml of Normal saline intraarticular injection to the knee joint weekly for 5 weeks
  Interventions: Drug: normal saline,2 ml., intraarticular weekly for 5 weeks
- A (Experimental): 2 ml of 25 mg sodium hyaluronate intraarticular injection to the knee joint weekly for 5 weeks
  Interventions: Drug: 25 mg sodium hyaluronate "GO ON"

INTERVENTIONS:
Drug: 25 mg sodium hyaluronate "GO ON" — 25 mg sodium hyaluronate, 2 ml., intraarticular weekly for 5 weeks
  Arms: A
Drug: normal saline,2 ml., intraarticular weekly for 5 weeks
  Arms: B

SUMMARY:
OA knee is a common degenerative diseases of the joint.

* There are many methods to treat this condition.
* Hyaluronic acid is one of the recomended treatment of OA knee.
* There is no any study on MRI change after injection hyaluronic acid.
* The Hypothesis is 25 mg of sodium hyaluronate (2.5 ml) would preserve the joint space in patient with osteoarthritis of the knee compared to placebo .

DETAILED DESCRIPTION:
This will be the phase III randomized, double-blind, placebo-controlled trial of 52 weeks duration designed to evaluate the efficacy of sodium hyaluronate to placebo (saline), in adult with OA of the knee joints. Randomization will be stratified by Kellgren-Lawrence(KL) grade (garde2 or 3), by subjects X-ray. A total of 60 subjects are planed for enrollment in this study. The study will be conducted over approximately 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Ambulatory non pregnant females and males 40-<80 years of age.
* Subjects who withdraw pain medication or nutritional supplements for symptom relief for OA hand for a total of at least 30 days before screening visit 0.
* Pain at or below 40 mm on a 100 mm VAS in the index knee joints.
* A documented diagnosis of OA of the knee joint, or meeting American College of Rheumatology (ACR) clinical criteria for classification of idiopathic (primary) OA for at least 6 months prior to screening.
* Subject has been documented radiographic evidence of OA of the knees from the screening Visit radiograph of grade 2 or 3 according to Kellgren and Lawrence Radiographic Grading.
* Subject has no any contraindication for MRI
* Subject is able to understand and complete pain/function, global arthritis evaluation, and health outcome assessment.

Exclusion Criteria:

* Subjects with history of hypersensitivity to hyaluronate.
* Subjects with skin lesion at the knee joint.
* A history of knee surgery within 6 months prior to screening V0.
* Significant prior injury to the knee joint within 12 months prior to screening V0.
* Disease of the spine or other lower extremity joints of sufficient degree to affect the knee joint.
* Treatment with other drugs potentially affecting bone or cartilage metabolism as described below:
* chronic systematic corticosteroids
* Diacerin or glucosamine treatment within the last 12 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
MRI will be analysed with semiquantitative whole organ scoring method (WORMS) c | 6 months

SECONDARY OUTCOMES:
WOMAC, VAS, side effects | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Weerachai Kosuwon, Professor, Principal Investigator — Faculty of Medicine, Khon Kaen University
Locations (1):
- Weerachai Kosuwon, Khon Kaen, Changwat Khon Kaen, Thailand